CLINICAL TRIAL: NCT05689125
Title: Bougies as Aid for Endotracheal Intubation Via Video Laryngoscopy During Continuous Chest Compressions by Anesthesia Residents: a Randomized Crossover Simulation Trial
Brief Title: Bougies as Aid for Endotracheal Intubation Via Video Laryngoscopy During Continuous Chest Compressions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Huang YuGuang, MD, Peking Union Medical College Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: K2562
Record Dates: First submitted 2023-01-06; First posted 2023-01-18 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Endotracheal Intubation; Cardiopulmonary Resuscitation; Simulation

STUDY DESIGN:
Intervention Model Description: Participants will perform endotracheal intubation by four methods in a randomized order. The four methods are endotracheal intubations assisted by a railroaded bougie, assisted by a preloaded bougie, assisted by a stylet, and with no assistance.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Railroaded bougie (Experimental): An endotracheal tube is loaded onto a bougie posterior to the placement of the bougie into the trachea.
  Interventions: Device: Railroaded bougie
- Preloaded bougie (Other): An endotracheal tube is loaded onto a bougie prior to initiating laryngoscopy.
  Interventions: Device: Preloaded bougie
- Stylet (Active Comparator): A stylet is placed within an endotracheal tube prior to initiating laryngoscopy.
  Interventions: Device: Stylet
- Naked endotracheal tube (No Intervention): Residents expose the glottis by a video laryngoscope and perform the endotracheal intubation without assistance of stylet or bougie.

INTERVENTIONS:
Device: Railroaded bougie — Residents expose the glottis by a video laryngoscope and place the tip of bougie through the vocal cords. Then, an assistant loads an endotracheal tube on the free end of the bougie. Residents advance the endotracheal tube over the bougie and withdraw the bougie.
  Arms: Railroaded bougie
Device: Preloaded bougie — Residents expose the glottis by a video laryngoscope and perform the endotracheal intubation using a bougie with a preloaded endotracheal tube while an assistant secures the free end of the bougie. Residents withdraw the bougie when the endotracheal tube reaches an appropriate depth.
  Arms: Preloaded bougie
Device: Stylet — Residents expose the glottis by a video laryngoscope and perform the endotracheal intubation with the assistance of a stylet. An assistant withdraws the stylet when the tip of the endotracheal tube passes through the vocal cords. Then residents place the endotracheal tube to an appropriate depth.
  Arms: Stylet

SUMMARY:
The goal of this clinical trials is to analyze the effects of using bougies as adjuncts on the performance of endotracheal intubation via video laryngoscopy during cardiopulmonary resuscitation in anesthesia residents. The main question it aims to answer is whether bougie use has a significant effect on first-attempt failure of endotracheal intubation via video laryngoscopy during continuous chest compressions. Participants will perform endotracheal intubation via video laryngoscopy by four methods in a randomized order in a simulated cardiopulmonary resuscitation scenario on a manikin. The four methods are endotracheal intubations assisted by a railroaded bougie, assisted by a preloaded bougie, assisted by a stylet, and with no assistance. Researchers will compare the first-attempt failure rate of the four methods to see if a railroaded bougie method has a significant different first-attempt failure from that of the other three methods.

ELIGIBILITY:
Inclusion Criteria:

* Residents who are enrolled in the three-year standardized residency training program in the Department of Anesthesiology, Peking Union Medical College Hospital in February, 2023.

Exclusion Criteria:

* Residents who refuse to participate and residents who fail the pre-test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2023-02-09 (Actual); Primary Completion 2023-02-20 (Actual); Study Completion 2023-02-20 (Actual)

PRIMARY OUTCOMES:
Failure on the first attempt | At the completion of the intubation
  An attempt is terminated and defined as a failure when a resident tries for one minute but is still unable to start ventilation, or when a resident feels unable to succeed and decides to give up, or when a resident withdraws a laryngoscope blade, a bougie, or a tube out of the month after the initial insertion. This outcome will be measured based on videos of endotracheal intubation procedures recorded by a camera placed on the right side of the manikin.

SECONDARY OUTCOMES:
Failure on two attempts | At the completion of the intubation
  If the first attempt of a method fails, the resident will be given a second opportunity of the same method. This outcome will be measured based on videos of endotracheal intubation procedures recorded by a camera placed on the right side of the manikin.
Duration of the first attempt | At the completion of the intubation
  The time elapsed between the insertion of a laryngoscope blade into the month and either the start of ventilation in a successful attempt or the termination of a failed attempt. This outcome will be measured based on videos of endotracheal intubation procedures recorded by a camera placed on the right side of the manikin.
Overall intubation duration | At the completion of the intubation
  Duration of the first attempt if it succeeds or the sum of the duration of both attempts if the first attempt fails. This outcome will be measured based on videos of endotracheal intubation procedures recorded by a camera placed on the right side of the manikin.
Self-reported intubation difficulty | At the completion of the intubation
  0-10 ranking scale with 0 representing "the easiest" and 10 "the most difficult" rated by the residents.

CONTACTS AND LOCATIONS:
Overall Officials: Xu Li, MD, Study Chair — Peking Union Medical College Hospital; Yuguang Huang, MD, Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
The study plan can be obtained from the principal investigator on request.

REFERENCES:
- [Derived] Xu X, Ma H, Zhang Y, Liu W, Jung B, Li X, Shen L. Efficacy of bougie first approach for endotracheal intubation with video laryngoscopy during continuous chest compression: a randomized crossover manikin trial. BMC Anesthesiol. 2024 May 21;24(1):181. doi: 10.1186/s12871-024-02560-3. PMID 38773386